CLINICAL TRIAL: NCT02286635
Title: A Phase 1, Open-Label, 2-Arm, Fixed-Sequence Study to Evaluate the Potential Effects of Multiple Doses of Rifampin (CYP3A4 Inducer) and Clarithromycin (CYP3A4 Inhibitor) on the Single Dose Pharmacokinetics of Deflazacort in Healthy Subjects
Brief Title: Evaluate Effects of Multiple Doses of Rifampin and Clarithromycin on the Single Dose Pharmacokinetics of Deflazacort
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-104-CL-025
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — deflazacort; Rifampin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A Deflazacort and Rifampin (Experimental): Subjects will recieve one 18 mg dose of deflazacort on Day 1, Period 1 and Day 10, Period 2; cohort A. Subjects will receive once daily dosing of rifampin on Day 1, Period 2 through Day 10, Period 2.
  Interventions: Drug: Deflazacort and rifampin
- Cohort B Deflazacort and Clarithromycin (Experimental): Subjects will recieve one 18 mg dose of deflazacort on Day 1, Period 1 and Day 4, period 2; cohort B. Subjects will receive twice daily dosing of clarithromycin on Day 1, Period 2 through Day 4, Period 2.
  Interventions: Drug: Deflazacort and Clarithromycin

INTERVENTIONS:
Drug: Deflazacort and rifampin — Deflazacort, a glucocorticoid with anti-inflammatory and immunosuppressive effects, is used in treating a variety of diseases. Pharmacologically it is an inactive pro-drug which is metabolized completely and rapidly to the active drug 21-desacetyldeflazacort (21 desacetyl-DFZ). The elimination of this metabolite is primarily via the urine in humans. Its potency is approximately 70 to 90% of prednisone and 6 mg of deflazacort has approximately the same anti-inflammatory potency as 5 mg of prednisolone or prednisone. Rifampin is a potent inducer of drug metabolism by inducing a variety of hepatic and intestinal CYP enzymes, especially CYP3A4. Rifampin is a semi-synthetic antibiotic.
  Other Names: DFZ
  Arms: Cohort A Deflazacort and Rifampin
Drug: Deflazacort and Clarithromycin — Deflazacort, a glucocorticoid with anti-inflammatory and immunosuppressive effects. It is an inactive pro-drug which is metabolized completely and rapidly to the active drug 21 desacetyl-DFZ. The elimination of this metabolite is primarily via the urine in humans. Its potency is approximately 70 to 90% of prednisone. Clarithromycin is a semi-synthetic macrolide antibiotic. Clarithromycin is active in vitro against a variety of aerobic and anaerobic gram-positive and gram-negative bacteria as well as most mycobacterium avium complex (MAC) bacteria. Additionally, the 14-OH clarithromycin metabolite also has clinically significant antimicrobial activity. Clarithromycin is indicated for the treatment of mild to moderate infections such as pharyngitis/tonsillitis.
  Other Names: biaxin
  Arms: Cohort B Deflazacort and Clarithromycin

SUMMARY:
The primary objective of the study is to determine the potential effects of multiple doses of rifampin and clarithromycin on the single dose pharmacokinetics (PK) of the deflazacort active metabolite (21 desacetyl-DFZ) in healthy adult subjects.

DETAILED DESCRIPTION:
This is an open label, parallel 2-arm, 2-period, fixed-sequence study in 58 healthy adult non-tobacco using male and female subjects divided into 2 cohorts, with 29 subjects in each arm of the study (Cohorts A and B).

Cohort A:

On Day 1 of Period 1 a single oral dose of deflazacort (Treatment A) will be administered followed by PK sampling for 24 hours for 21 desacetyl DFZ and, if data permit, deflazacort.

In Period 2, multiple oral doses of rifampin will be administered once daily (QD) for 10 consecutive days with a single oral dose of deflazacort coadministered on Day 10 (Treatment B). Pharmacokinetic sampling for 21-desacetyl-DFZ and, if data permit, deflazacort will be taken for 24 hours following deflazacort dosing on Day 10. Morning urine collection will be used to measure 6β-hydroxycortisol and free cortisol concentrations on Days 1, 4, 8, and 10 to evaluate the level of cytochrome P450 (CYP) enzyme induction.

Cohort B:

On Day 1 of Period 1 a single oral dose of deflazacort (Treatment C) will be administered followed by PK sampling for 24 hours for 21-desacetyl-DFZ and, if data permit, deflazacort.

In Period 2, multiple oral doses of clarithromycin will be administered twice daily (BID) for 4 consecutive days with a single oral dose of deflazacort coadministered on the morning of Day 4 (Treatment D). Pharmacokinetic sampling for 21 desacetyl-DFZ and, if data permit, deflazacort will be taken for 24 hours following deflazacort dosing on Day 4.

Both Cohorts A and B:

There will be at least 24 hours between the dose in Period 1 and the first dose in Period 2.

Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

The clinic will attempt to contact subjects using their standard procedures approximately 14 days after the last study drug administration to determine if any adverse events (AEs) have occurred since the last dose of study drug. Subjects who terminate the study early will be contacted if the Principal Investigator (PI) deems necessary.

Cohort A:

Treatments A and B are described as follows:

Treatment A (Period 1): 18 mg deflazacort (3 x 6 mg tablets) at Hour 0 on Day 1, following an overnight fast.

Treatment B (Period 2): 600 mg rifampin (2 x 300 mg capsules) administered at Hour 0 after an overnight fast every 24 hours for 10 days (within ± 1 hour of dosing time on Day 1), with 18 mg deflazacort (3 x 6 mg tablets) coadministered on Day 10.

Cohort B:

Treatments C and D are described as follows:

Treatment C (Period 1): 18 mg deflazacort (3 x 6 mg tablets) at Hour 0 on Day 1, following an overnight fast.

Treatment D (Period 2): 500 mg clarithromycin (1 x 500 mg tablets) administered at Hour 0 and Hour 12, under fasting conditions, approximately every 12 hours, for 4 days (within ± 1 hour of dosing times on Day 1), with 18 mg deflazacort (3 x 6 mg tablets) coadministered at Hour 0 on the morning of Day 4. The final dose of clarithromycin will be given at Hour 12 in the evening of Day 4.

All study drugs in both cohorts will be administered orally with approximately 240 mL of water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, 18 55 years of age
* Continuous non smoker who has not used nicotine containing products for at least 3 months
* Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2
* For a female of non childbearing potential: must have undergone a sterilization procedures or be postmenopausal with amenorrhea for at least 1 year prior to the first dose of study drug and FSH serum levels consistent with postmenopausal status
* A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days
* If male, must agree not to donate sperm from the first dose of study drug until 90 days

Exclusion Criteria:

* Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
* History or presence of alcoholism or drug abuse within the past 2 years
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds (e.g., steroids or their formulations including lactose)
* History or presence of:

  1. Symptomatic cardiomyopathy at screening
  2. Immunosuppression or other contraindications for corticosteroid treatment
  3. History of chronic systemic fungal or viral infections
  4. Galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption
  5. Diabetes mellitus
  6. Osteoporosis
  7. Myasthenia gravis
  8. Epilepsy
  9. Idiopathic hypocalcuria
  10. Hypothyroidism (TSH clinically significant)
  11. Gastrointestinal issues or ulcers
  12. Previous corticoids-induced myopathy
  13. Ocular herpes simplex
* Female subjects of childbearing potential
* Female subjects who are pregnant or lactating
* Positive urine drug or alcohol results
* Positive urine cotinine
* Positive results for HIV, HBsAg or HCV
* Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg
* Seated heart rate is lower than 40 bpm or higher than 99 bpm
* QTc interval is > 430 msec (males) or > 450 msec (females)
* Has received any live or live-attenuated vaccine within 30 days
* Has received any immunosuppressive agents, coal tar, and/or radiation therapies within 30 days
* Has received injectable corticoids in the 12 weeks dose of study drug or any oral form of corticoids in 30 days
* Estimated creatinine clearance < 80 ml/min
* Unable to refrain from or anticipates the use of

  * Any drug, including prescription and non prescription medications, as well as herbal remedies known to be significant inhibitors of CYP 3A4 enzymes and/or P gp for 14 days
  * Any drugs known to be significant inducers of CYP 3A4 enzymes and/or P gp, including St. John's Wort, for 28 days
* Have been on a diet incompatible with the on study diet within 28 days
* Donation of blood or significant blood loss within 56 days
* Plasma donation within 7 days
* Participation in another clinical trial within 28 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effects of CYP3A4 inhibitors and inducers on the pharmacokinetics (PK) of deflazacort in healthy subjects including the area under the plasma concentration time curve, from time 0 to the last measurable non-zero concentration. | 10 days and 4 days
  Effects of CYP3A4 inhibitors and inducers on the pharmacokinetics (PK) of deflazacort in healthy subjects including the area under the plasma concentration time curve, from time 0 to the last measurable non-zero concentration.

SECONDARY OUTCOMES:
Safety and tolerability of one dose of deflazacort in healthy subjects receiving CYP3A4 inhibitors and inducers as measured by capturing occurrence of adverse events. | 10 days and 4 days
  Safety and tolerability of one dose of deflazacort in healthy subjects receiving CYP3A4 inhibitors and inducers as measured by capturing occurrence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bioscience Center, Study Director — Marathon Pharmaceuticals, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States